CLINICAL TRIAL: NCT01944735
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CTX-4430 When Administered Orally to Cystic Fibrosis Patients for Fifteen Days
Brief Title: Phase 1 Study Assessing the Safety and Tolerability of CTX-4430 in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celtaxsys, Inc. (Other)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTX-4430-CF-001
Record Dates: First submitted 2013-09-06; First posted 2013-09-18 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — acebilustat; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Once daily oral capsule containing 50 or 100 mg of CTX-4430
  Interventions: Drug: CTX-4430
- Placebo (Placebo Comparator): Once daily oral capsule containing mannitol, visibly identical to CTX-4430 capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CTX-4430 — Ascending repeat doses of CTX-4430 will be administered orally, once-daily, to patients in 2 cohorts on days 1-15.
  Arms: Active
Drug: Placebo — Repeat doses of placebo will be administered orally, once-daily, to patients in 2 cohorts on days 1-15
  Other Names: Mannitol
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of multiple oral doses of CTX-4430 when administered to cystic fibrosis (CF) patients once-daily (QD) for 15 days.This study will include two dose levels. For each dose level, blood samples will be collected for exploratory PK and PD assay validation. In addition, sputum will be collected for exploratory biomarker analysis. Following multiple dose administration, pulmonary function and exploratory lung clearance index (LCI) measurements will be taken.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, 18 to 55 years of age (inclusive) at the time of screening.
2. Confirmed diagnosis of CF based on the following: positive sweat chloride or sodium value ≥ 60 mEq/L, and/or genotype with two identifiable mutations consistent with CF, accompanied by one or more clinical features consistent with the CF phenotype or a diagnosis of CF made by a specialist in this condition.
3. In the judgment of the Principal Investigator (PI), the patient is medically stable with no change in symptoms, medication, or with clinical laboratory results that in PI opinion are compatible with the diagnosis of either CF or a complication thereof and are judged acceptable for inclusion.
4. Body mass index (BMI) ≥ 17.0 (kg/m2).
5. Non-tobacco/nicotine-containing product user for a minimum of 6 months prior to the first study drug administration.
6. Forced Expiratory Volume (FEV1) of >50% and <90% of predicted at screening.
7. Must agree to use adequate method of contraception.

Exclusion Criteria:

1. Patient has displayed any significant clinical/laboratory/radiological/spirometric sign of unstable or unexpectedly deteriorating respiratory disease within 30 days prior to the first study drug administration.
2. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease that depart from the patient's usual baseline level of health as a patient with CF.
3. Has a history of lung transplantation.
4. History or presence of alcoholism or drug abuse within 2 years prior to the first study drug administration.
5. Personal or family history of prolonged QT syndrome; or a QTc interval >430 msec (males) or >450 msec (females) using Bazett's formula (QTcB) or deemed clinically significant by the PI.
6. Sitting blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg, unless deemed clinically insignificant by the PI.
7. Pulse is higher than 100 b.p.m or lower than 50 b.p.m. unless deemed clinically insignificant by the PI.
8. Failure to satisfy the PI of fitness to participate for any other reason.
9. In the judgment of the PI, clinically significant hemoptysis (>30 cc per episode) within the last 180 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and tolerability of multiple oral doses of CTX-4430 when administered to cystic fibrosis (CF) patients once-daily (QD) | 15 days
  Changes in clinical signs and symptoms of safety data that include physical examinations, ECGs, vital signs, pulse oximetry, pulmonary function (spirometry), clinical laboratory results, and adverse events which will be summarized descriptively and reported in tabular form.

CONTACTS AND LOCATIONS:
Overall Officials: J Stuart Elborn, MD, FRCP, Principal Investigator — Queen's University, Belfast
Locations (4):
- United Kingdom (4):
  - The Medicinces Evaluation Unit, Wythenshawe, Manchester
  - Celerion, Belfast, Northern Ireland
  - Glasgow Clinical Research Facility, Glasgow
  - Royal Brompton Hospital, London